# EFFECT OF PROPOLIS PASTE AS INTRACANAL MEDICAMENT ON POST-ENDODONTIC PAIN: A DOUBLE BLIND RANDOMIZED CLINICAL TRIAL

#### **SYNOPSIS**

Approved by the Scientific Committee
Approved by Institutional Review Board
Approved by Board of Advanced Studies and Research
Trial registered with ISRCTN (Biomed Central) – ISRCTN66816132
Dow University of Health Sciences
In partial fulfillment of the requirement
For the Degree of

**Masters in Dental Surgery** 

Ву

Dr. Juzer Shabbir Saifee



Dr. Ishrat-ul-Ibad Khan Institute of Oral Health Sciences

**Dow University of Health Sciences** 

Karachi, Pakistan

14 November, 2017

**CORRESPONDING SUPERVISOR:** 

Dr. Fazal-ur-Rehman Qazi

#### CERTIFICATE

#### Researcher (first author):

Name:

Dr. Juzer Shabbir Saifee

Designation: M.D.S. Trainee

Department: Operative Dentistry

Qualification: B.D.S., M.D.S trainee

Signature:

#### Supervisor (corresponding author):

Dr. Fazal-ur-Rehman Qazi

Designation: M.D.S Program Director, Associate Professor.

Department: Operative Dentistry

Qualification: B.D.S., F.C.P.S.

Signature:

2

### **TABLE OF CONTENTS**

| TITIE | 1 |
|--------------------------------------|----|
| Certificate | 2 |
| Contents | 3 |
| ABSTRACT | 4 |
| CHAPTER 1: INTRODUCTION | |
| 1.1. Background | 6 |
| 1.2. Literature Review | 8 |
| 1.3. Rationale of Study | 10 |
| 1.4. Statement of Problem | 10 |
| 1.5. Objectives | 11 |
| 1.6. Hypothesis | 11 |
| 1.7. Operational Definitions | 11 |
| CHAPTER 2: METHODOLOGY | |
| 2.1. Study Design | 13 |
| 2.2. Study Setting | 13 |
| 2.3. Study Duration | 13 |
| 2.4. Study Population | 13 |
| 2.5. Sample Size | 14 |
| 2.6. Sampling Technique | 15 |
| 2.7. Data Collection Procedure | 16 |
| 2.8. Study Variables | 17 |
| 2.9. Statistical Analysis | 18 |
| CHAPTER 3: REFERENCES AND APPENDICES | 19 |

#### <u>ABSTRACT</u>

#### **Background:**

Dental pain is a significant factor due to which the patient seeks treatment. Non-surgical Endodontic treatment is a major therapy to treat the pain and save the tooth. Pain control during this endodontic procedure is a challenging goal for dental practitioners. Patients having necrotic teeth have the highest incidence of post-endodontic pain, therefore, it needs special attention.

To prevent post-endodontic pain, different techniques have been adapted. Placing biocompatible medications having either potent antimicrobial activity or anti-inflammatory component or both inside the root canals is one of the eminent techniques to disinfect the canals and control the pain. Calcium hydroxide is the most common intracanal medicament to which all other medicaments are being compared but it carries certain drawbacks with it. It is ineffective against E.faecalis and Fungi, lacks anti-inflammatory component and is controversial in preventing pain. Presently, focus of research has shifted towards natural alternatives to synthetic intracanal medication. Propolis is an organic resinous substance obtained from bee hive. It is nontoxic, biocompatible, anti-inflammatory, anti-oxidant, and anti-microbial and is effective against E.faecalis and fungi.

#### **Objective:**

To evaluate the effect of Propolis paste on post-endodontic pain in comparison to calcium hydroxide at different time intervals.

#### **Trial Design:**

A parallel group prospective double blind randomized control (clinical) trial.

#### **Methods:**

This study will be conducted in Department of Endodontics, Dow International Dental College within

year after approval. 80 patients having painful, single rooted necrotic teeth with PAI index 3

and 4 will be selected and randomly assigned to either control (Group I) or experimental (Group II).

Randomization will be computer generated and the produced sequence will be placed in sealed envelope

with allocation concealment from the principal researcher. Patients will be blinded to group assignment and the principal researcher will be blinded from the type of intracanal medicament being inserted. Standard non-surgical endodontic procedure will be performed by the principal researcher till root canal preparation is completed. Intracanal medicaments will then be inserted by a secondary operator in the first visit. In Group I, calcium hydroxide will be inserted. In group II (experimental), Propolis powder mixed with saline will be inserted. Visual Analogue Pain Scale will be provided to the patients to rate their pain intensity pre-operatively, then at 4 hours, 12 hours, 24 hours, 48 hours and 72 hours after treatment. Visual analogue scales will be collected after 4 days.

#### **Statistical Analysis:**

Analysis of the data will be done through IBM SPSS v24. Flare-up will be identified as increase of 20 or more points on Visual analogue scale from initial pain score. Repeated Measure ANOVA will be used to compare pain scores between the groups at various time intervals; Mann-Whitney U test will be applied for comparison of pain between gender; and Kruskal-Willis test will be applied for comparison of pain between age groups. Crosstabs will be used to report the rate of flare-up.

#### **Key words:**

Propolis, Calcium hydroxide, Pain, Flare up, Intracanal Medications, Necrotic teeth.

#### **CHAPTER 1: INTRODUCTION**

#### 1.1 - Background:

Dental Pain is a significant factor, due to which the patient seeks treatment and endodontic therapy is a major treatment to alleviate the pain<sup>(1)</sup>. The occurrence of mild pain after root canal preparation is not uncommon<sup>(2)</sup>. But sometimes, endodontic procedure can result in flare-up. Flare up can be defined as severe pain and/or swelling of the area of endodontically treated tooth occurring within few hours to few days following initiation and/or completion of root canal treatment<sup>(3)</sup>. Severe post-endodontic pain is an emergency, which requires a prompt intervention. Failure to control the post endodontic pain results in demotivation of the patient and eventual extraction of the affected tooth.

The cause of post-endodontic pain is the peri-radicular inflammation which results due to extrusion of irritants from the root canals into the periapical region<sup>(3)</sup>. These irritants might be of nonmicrobiological and microbiological origin<sup>(4)</sup>. Non-microbiological cause is mainly due to iatrogenic errors; inaccurate working length estimation, in-correct method of root canal preparation, overinstrumentation and extrusion of obturating materials, intracanal medicaments and chemical irrigants<sup>(3)</sup>. These iatrogenic errors can be controlled by carefully performing endodontic procedures. But sometimes, even after careful and judicious endodontic procedure, flare up occurs, which is due to microbiological cause<sup>(5)</sup>. The microbiological factor is the most common cause of peri-radicular inflammation. It includes the apical extrusion of infected debris, changes in endodontic microbiota or in environmental conditions, secondary intra-radicular infection and increase in oxidation-reduction potential<sup>(5)</sup>. The Bacteria which are predominant in symptomatic apical periodontitis are Parvimonas micra, Eubacterium, Porphyromonas and Prevotella<sup>(3)</sup>. Many chemical mediators are responsible for the occurrence of pain during inflammation. Few examples are; histamine, serotonin, prostaglandins, platelet activating factors and leukotrienes. Certain plasma mediators are also directly or indirectly involved in induction of pain, like; Hageman factor, Bradykinin and fibrinopeptides<sup>(6)</sup>.

In some studies, the incidence of flare-up is found to be upto 50% <sup>(7-9)</sup>. According to a systemic review, mean post-treatment pain prevalence at 24 hours is 40%. Moreover, moderate pain severity was reported to be 24% at 24 hours<sup>(1)</sup>. In a meta-analysis, frequency of flare-up was found to be 8.4%

(10).

Management of flare up includes prescribing analgesics and antibiotics, performing occlusal reduction, re-instrumentation, placing of intracanal medications, incision and drainage, and cortical trephination <sup>(11)</sup>. Although, chemo-mechanical preparation using sodium hypochlorite irrigation is of paramount importance for reduction of bacterial load in root canals, but 40-60% of the canals still remain infected with pathogenic bacteria<sup>(12-14)</sup>. Intracanal medicaments are recommended to supplement the chemo-mechanical preparation and eliminate the persistent bacteria in the root canal system <sup>(14, 15)</sup>.

According to Walton<sup>(16)</sup>, The role of intracanal medicament is to; eliminate the microbes, render canal contents inert, control persistent periapical abscesses, prevent or control post-treatment pain and enhance anesthesia. The most commonly used intracanal medicament is Calcium hydroxide<sup>(2)</sup>. Incomplete elimination of gram-negative bacteria, questionable healing of periapical lesions and inept elimination and prevention of post-endodontic pain <sup>(2, 4, 17)</sup> are some limitations of using calcium hydroxide. Intracanal use of corticosteroid and antibiotic containing medication like ledermix paste has been found to be effective to control the post-endodontic pain<sup>(8)</sup>. But, yeasts are resistant to it<sup>(18)</sup> and ledermix paste is associated with discoloration of tooth<sup>(19)</sup>. Also, it has been found to have a potential to cause increased degree of inflammation <sup>(20)</sup>. More recently trends have shifted towards finding a natural organic alternative <sup>(21)</sup> to synthetic inorganic intracanal medicaments. Propolis is a natural product which has been used extensively in past<sup>(22)</sup>. It has anti-microbial and antiinflammatory properties and can be used as an intracanal medicament for disinfection of the root canal system<sup>(23)</sup>. Propolis is found to be effective against E.faecalis, S. aureus and C.albicans and other endodontic pathogens <sup>(24-26)</sup>. It is also effective against some gram-negative bacteria<sup>(27)</sup>. Propolis also decreases

Lipopolysaccharide(LPS) induced inflammation<sup>(28)</sup>. Although no harmful effect of propolis has been reported till date, the only drawback of propolis found is its potential to cause

allergic contact dermatitis (29-31).

As microbes are the most common cause of post endodontic pain, the incidence of post endodontic pain is reduced when intracanal medicaments are used for disinfection<sup>(5)</sup>. Furthermore, several studies have shown that components of Intracanal medicaments are able to diffuse through dentinal tubules, ramifications and apical foramen to exert their effect in inaccessible areas inside the tooth and periapical area <sup>(32-38)</sup>. Owing to the fact that Propolis is effective against endodontic pathogens and has anti-inflammatory component; flavonoid<sup>(39)</sup>, it is expected to reduce the occurrence and severity of postendodontic pain in necrotic teeth. The aim of the present study is to test the clinical efficacy of propolis when used as intracanal medicament in reducing and preventing the post-endodontic pain as compared to calcium hydroxide.

#### 1.2 - Literature Review:

As the non-surgical endodontics is developing, there have been significant development in prevention and treatment of post-endodontic pain but controversy remains on the effectiveness of the intracanal medicaments in reducing pain<sup>(3)</sup>. There is also no systemic review or meta-analysis published till date about the role of intracanal medicament in prevention of post-endodontic pain.

Calcium hydroxide has been broadly used for various purposes in dentistry since 1920s. Today, it is still the most widely used endodontic medicament all over the world<sup>(40)</sup>. The mechanism of action by which calcium hydroxide kills the bacteria is related to its high pH. The micro-organisms are killed due to release of hydroxyl ions, which results in highly alkaline environment in which bacteria are unable to survive<sup>(41)</sup>. Calcium hydroxide has also shown to inactivate bacterial lipopolysaccharide (LPS) and assist in periapical tissue healing<sup>(42)</sup>. In few studies, calcium hydroxide has been reported to be useful in controlling inflammatory exudate from peri-radicular region. Mechanism behind this property might be related to its antimicrobial effect<sup>(43)</sup>, capillary contraction<sup>(44)</sup> and apical plug formation<sup>(43)</sup>. Clinically, it was suggested that calcium hydroxide had pain-relieving property due to its

antibacterial and tissue altering effects<sup>(45)</sup>. But some authors have disagreed with this suggestion and reasoned that calcium hydroxide could initiate or increase pain by starting or exacerbating inflammation<sup>(46)</sup>. Likewise, few studies have shown that calcium hydroxide has no impact on prevention or reduction of post endodontic pain <sup>(47-50)</sup>.

Propolis is a byproduct, prepared by honey bees which has broad spectrum of biological activities<sup>(51)</sup>. Raw propolis consists of 50% plant resins, 30% waxes, 10% aromatic and essential oils, 5% pollens and 5% other organic substances<sup>(39)</sup>. Propolis has been found to be effective in treating colds, wounds and ulcers, sprains, rheumatism, heart disease, diabetes<sup>(52-55)</sup> and dental caries<sup>(56-60)</sup> due to its antiinflammatory<sup>(55, 61-63)</sup>, anti-microbial, anti-oxidant, anti-tumor<sup>(64)</sup>, anti-ulcer and anti-HIV properties<sup>(65)</sup>. The main constituents of temperate climate region propolis are flavonoids without Bring substituents, like chrysin, Galangin, pinocembrin and pinobanksin<sup>(39)</sup>. Being a major component of propolis, flavonoids are greatly responsible for pharmacological activities of it.

Several studies have been conducted regarding potential use of propolis in dentistry. Some studies have shown that propolis is effective in preventing and treating gingival and periodontal disease <sup>(66-69)</sup>. Propolis also has antiviral effects and can be used locally in viral infections<sup>(70)</sup>. Propolis is extremely effective medium for avulsed tooth <sup>(71-73)</sup>. Local application of propolis assist in healing wounds after oral surgery procedures, reduces inflammation and has analgesic effect<sup>(74, 75)</sup>. Propolis has a positive effect on bone forming during expansion of palatine suture<sup>(76)</sup>. It can reduce dentinal hypersensitivity by partially impregnating the tubules<sup>(77)</sup>. Propolis can also be used effectively as a direct pulp capping agent <sup>(78-80)</sup>.

There are several in-vitro studies regarding the use of propolis in endodontics. In few studies, it has been shown that Propolis can eliminate E.faecalis and C.albicans and reduce endotoxin when used as an intracanal irrigant<sup>(81,82)</sup>. In some studies, propolis was found to be more effective than calcium hydroxide against endodontic pathogens when used as an intracanal medicament <sup>(83,84)</sup>. Furthermore, propolis has also been found to be superior to tri-antibiotic mixture against E.faecalis<sup>(85)</sup>. Although, few studies have shown that chlorhexidine is more effective against E.faecalis as compared to propolis<sup>(83)</sup>.

<sup>86)</sup>. One study has shown that effectiveness of propolis is similar to chlorhexidine at 7 days<sup>(87)</sup>. Regarding the biocompatibility and toxicity, propolis has been found to be least toxic and highly biocompatible as compared to other endodontic medicaments and materials <sup>(78, 88-91)</sup>. The mechanism by which propolis induces its anti-inflammatory and analgesic action is through suppression of LPS-induced inflammatory response of key cells<sup>(92)</sup>. Yet, there is no in-vivo study performed to show the efficacy of propolis paste in reducing inter-appointment pain.

#### 1.3 - Rationale Of Study:

Necrotic teeth require an intracanal medicament which can effectively eliminate notorious bacteria and their byproducts from root canal system and thereby decrease chances of flare up and inter appointment pain indirectly by banishing the cause. Secondly, in order to eliminate and prevent pain and inflammation directly, an intracanal medicament must have an anti-inflammatory component in it. Calcium hydroxide has been proved to be ineffective against some of the detrimental endodontic pathogens and lacks anti-inflammatory component. To offset the draw back of a single intracanal medicament, two or more medicaments are mixed together which increases the cost. Propolis is a natural product which is effective against resistant microbes, is anti-inflammatory and cheaper than other synthetic medicaments. The literature lacks an in-vivo study that investigates the role of Propolis on post-endodontic pain. This study will be an attempt to fill this knowledge gap.

#### 1.4 - Statement Of The Problem:

Do propolis paste have any significantly better effect on preventing and eliminating the postendodontic pain as compared to calcium hydroxide?

#### 1.5 - Objectives:

To evaluate the effect of Propolis paste on post-endodontic pain in comparison to calcium hydroxide at different time intervals.

#### 1.6 - Hypothesis:

*Null hypothesis* ( $H_0$ ) = There will be no significant difference between Calcium hydroxide and Propolis paste in reducing and preventing post-endodontic pain.

Alternative hypothesis  $(H_A)$  = There will be a significant difference between Calcium hydroxide and Propolis paste group in reducing and preventing post-endodontic pain.

#### 1.7 - Operational Definitions:

#### Necrotic teeth:

The teeth which are tender to vertical percussion, have visible periapical widening or radiolucency on periapical radiograph without bone expansion (PAI index= 3 and 4) and shows no bleeding when the pulp chamber is opened.

#### PAI index (93):

- 1-Normal Periapical structure
- 2-Small changes in bone structure not pathognomic of apical periodontitis
- 3-Changes in bone structure with some mineral loss characteristic of apical periodontitis
- 4-Periodontitis with well-defined radiolucency
- 5-Severe periodontitis with exacerbating features and bone expansion.

#### VAS scale (94):

- No pain= Pain score 0.
- Mild pain intensity with no requirement of analgesics= Pain score 1-24.
- Moderate pain intensity with requirement of ibuprofen or similar medication= Pain score 25 –
   49.

- Severe pain intensity with requirement of narcotic analgesic= Pain score 50 74.
- Extreme pain intensity, not relieved by any type of medication= Pain score 75 100.

#### Flare-up:

An increase of 20 or more points from initial intensity of pain on Visual Analogue Scale (VAS)<sup>(94)</sup>.

#### **CHAPTER 2: METHODOLOGY**

#### 2.1 - Study Design:

The study will be a parallel group prospective double blind randomized controlled trial, with equal randomization (1:1). The patients and the principal researcher will be blinded from the type of intracanal medicament inserted.

#### 2.2 - Study Setting:

The study will be a multi-center research. It will be conducted in a secondary healthcare center; outpatient department of operative dentistry/endodontics in institutes / campuses of D.U.H.S, Karachi, Pakistan. It is a major commercial city of Pakistan having population of over 23.5 million<sup>(95)</sup>.

#### 2.3 - Study Duration:

One year.

#### 2.4 - Study Population:

Adults (aged 20 – 40) *Inclusion* 

#### criteria:

- Single rooted Necrotic teeth with symptomatic or aysmptomatic periapical periodontitis having visible periapical widening or radiolucency without bone expansion (PAI index 3 and 4).
- Teeth with favorable root morphology.
- Teeth with closed apex.

#### Exclusion criteria:

- Teeth with PAI index 1, 4 and 5.
- Patients who are on antibiotics.
- Patient with recent trauma to the jaw.

- Teeth with open apex
- Multi-rooted teeth.
- Vital teeth.
- Non-restorable teeth.
- Unfavorable root morphology (severely curved, dilacerated, severely sclerosed or obliterated).
- Teeth associated with soft tissue abscess or swelling.
- Teeth with external and internal root resorption
- Re-treatment cases.
- Periodontally compromised teeth (like mobile teeth and teeth with excessive bone loss).
- Teeth requiring endodontic surgery.
- Teeth requiring non-surgical endodontic treatment of multiple teeth in the same or opposing quadrant.
- Medically compromised patients (ASA-III and above), patients with special communication needs or who doesn't understand urdu or English language.
- Patients allergic to bee pollen or honey products.

#### 2.5 - Sample size:

Sample size was calculated using "Openepi" website, with following configuration:

- 90% power of the test
- 95% confidence interval (CI)
- With mean and standard deviation (SD) of Calcium hydroxide (2.42  $\pm$  2.1) and Creosote (1.12  $\pm$  0.66) from the article<sup>(96)</sup>.

The calculated minimum sample size was 62 (31 per group). We intended to increase sample size up to 30% Hence, final sample size was 80 (40 in each group).

#### 2.6 - Sampling technique:

Simple Random sampling technique will be used. Random allocation will be generated by computer with the help of independent person, not related to the study. Allocation concealment will be done by placing the sequence in sealed envelope by the independent person. The envelope will be given to the dental assistant not related to the study. After canal preparation is completed, the dental assistant will inform the secondary operator about which medicament to be inserted according to the sequence.

#### Details about primary operator:

Primary operator / principal researcher will be responsible for taking the written consent from the patients, diagnosis, selection of patients according to inclusion criteria and carrying out the endodontic procedure till the root canal preparation was completed. He will be blinded from the type of the medicament inserted into the root canal by the secondary operator. The primary operator / principal researcher will have an experience of 4 years of post-graduate training in the field of endodontics, with a total clinical experience of at least 6 years. The primary operator will also be responsible for; explaining the VAS scale to the patient, collecting the scale and data processing.

#### Details about secondary operator:

The secondary operator will be responsible for inserting the medicaments into the root canals after root canal preparation wi completed by primary operator. He will have an experience of 4 years of post-graduate training in the field of endodontics, with a clinical experience of at least 10 years. Additionally, the secondary operator will be given the training of mixing and inserting the medicaments into the root canals by Principal investigator for a week on a plastic block, resembling canal of a single rooted tooth (simulated canal block). The purpose of giving training on a plastic block is that the insertion of the medicaments can easily be observed according to its length and density achieved.

#### 2.7 - Data Collection Procedure:

Approval from Ethics Review Board will be obtained for this research. Written informed consent will be taken from patients.

The patients presenting in the Department of Endodontics will be included in the study according to inclusion criteria. Detailed medical and dental history will be obtained. Complete extra-oral and intraoral examination will be done and periapical radiograph will be taken. Diagnosis of the necrotic pulp with symptomatic or asymptomatic apical periodontitis will be made by the combination of history of pain, positive vertical percussion test (tender to percussion), Vitality test, periapical radiograph (having visible periapical widening or radiolucency) and no bleeding on opening of the pulp chamber.

The treatment will be performed by the principal researcher till the root canal preparation is completed. He will be blinded from the type of medicament being inserted by a secondary independent operator. In first visit, anesthesia (2% lidocaine, 1.8 ml with 1:100,000 epinephrine. Medicaine Inj.) will be given, rubber dam will be applied and standard infection control protocol will be followed<sup>(97)</sup>. Chamber will be opened with a sterilized round bur (ISO 001/014, BR-41. Mani,inc, Japan) and extension and refinement will be done with straight fissure bur(ISO 110/014, SF21.Mani,inc. Japan). After Chamber opening, glide path will be formed with ISO k file size 06, 08 and 10(Mani, Inc. Japan). Working length will then be taken with apex locator (Dentaport ZX. J Morita MFG Corp, Japan) and confirmed with radiograph. The preparation will be carried out till manual 20k hand file. Further canal preparation will be done in a crown down manner and rotary endodontic file system (Protaper universal, .04 taper. Dentsply Maillefer, Switzerland) will be used with the recommended torque (3.5 N) and speed (300 rpm). Ethylenediamine tetra acetic acid (EDTA) (GlydeFile prep, Dentsply Maillefer, Switzerland) will be used for lubrication and chelation during canal preparation. After each file introduced into the canal, irrigation will be done with 2.5% Sodium hypochlorite with a disposable, open ended, beveled, 27guage needle with 5ml syringe kept 2 mm short of working length and solution expressed in a slow passive manner. After canal preparation is completed, root canals will be irrigated with 10 ml sterile saline solution and then flooded with 17% EDTA solution (MD-Cleanser, Meta Biomed, Korea) for 3 mins to neutralize sodium hypochlorite. Then, the final rinse of 5 ml saline solution will be carried out (98). Canals will be dried with sterile paper points (Dentsply Maillefer, Switzerland) corresponding to master apical file.

Patients will be randomly divided into 2 groups of 40 patients each, according to the intracanal medication inserted. The type of medicament to be placed will be informed to the secondary operator by a dental assistant through computer generated sequence, who will insert the assigned intracanal medicament. Group I (control [treatment as usual]) will consist of teeth in which Calcium Hydroxide paste (Calcipulpe, Septodont. France) will be inserted. In Group II (experimental), 95% propolis powder (Henan Fumei Bio-technology Co., Ltd. China reg no.: 411082100010933) mixed with saline in a ratio of 1:1.5(wt/vol) to form paste, will be inserted into the root canals. These medicaments will be inserted into the canal with lentulo-spiral (Dentsply Maillefer, Switzerland) one size smaller than the master apical file, keeping it 1 mm short from the actual working length. Sterilized dry cotton wool will be placed in pulp chamber after insertion of medicaments and cavity will be filled with temporary cement (Cavit. ESPE Dental AG, Seefeld, Germany). Patient will be given a Visual (pain) analogue scale to rate their pain score. Patients will have to mark their intensity of pain preoperatively, then at different time intervals; 4 hours, 12 hours, 24 hours(day 2), 48 hours(day 3), 72 hours(day 4). Patients will be recalled after 7 days, visual analogue scale will be collected and data will be processed. Obturation and core build-up will be done after 7 days.

#### 2.8 - Study Variables:

- Dependent variable: pain score.
- Independent variable: gender, age, Necrotic teeth with PAI index 3 or greater

#### 2.9 - Statistical Analysis:

For data entry and analysis, IBM SPSS version 24 was used. For comparison of the mean pain scores between and within both the groups (Control and Experimental), repeated measure anova (mixed way anova) will be employed. Additionally, we will treat pain scores of patients taking pain killers (having pain scores of 25 or above) as missing values and the same analysis will be done; and a separate table will be reported for it. For multiple comparisons between and within groups, post hoc (LSD) test will be applied. For each group, descriptive statistics will be reported like mean, SD, minimum and

maximum of VAS pain scores. Furthermore, using mean pain scores of these tables, a line chart will be used to show the pain score trend with passage of time.

For comparison of pain score averages between the genders, Mann-Whitney U test will be applied.

Patients will be divided into four groups according to their ages; 20 to 24, 25 to 29, 30 to 34 and 35 to 40. For comparison of pain averages among the age groups, Kruskal Wallis test will be applied.

A p-value of 0.05 or less will be considered as significant and 0.01 or less as highly significant.

Descriptive statistics like frequencies will be used to report the statistics of: age (with percentages, mean age, SD, minimum and maximum); pre-operative pain status of sample; and the percentages of each type of single rooted teeth included in the study.

Similarly, the descriptive statistics like crosstabs will be used to analyze and report; the distribution of total number of males and females in each group; distribution of age groups in each group; the percentages of type of oral analgesics used by the patients according to different time intervals; the severity of pain experienced according to gender at different time intervals; and the severity of pain experienced by the patients according to age groups at different time intervals. Furthermore, the crosstab will also used to report flare-up rate according to each group. The flare-up will be determined as having pain score difference of 20 or more from previous time interval to the next one.

#### **CHAPTER 3: REFERENCES AND APPENDICES:**

#### 3.1 – References:

- 1. Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011;37(4):429-38.
- 2. Gama TG, de Oliveira JCM, Abad EC, Rôças IN, Siqueira Jr JF. Postoperative pain following the use of two different intracanal medications. Clin Oral Investig. 2008;12(4):325-30.
- 3. Sipavičiūtė E MR. Pain and flare-up after endodontic treatment procedures. Stomatologija. 2014;16:25-30.
- 4. Siqueira J, Barnett F. Interappointment pain: mechanisms, diagnosis, and treatment. Endod Topics. 2004;7(1):93-109.
- 5. Siqueira JF, Jr. Microbial causes of endodontic flare-ups. Int Endod J. 2003;36(7):453-63.
- Mittal R. Endodontic flare—ups: an overview. J Oral Health Comm Dent. 2010;4(3):67-71.
- 7. Christopher U, Emmanuel A. Flare-up incidence and related factors in adults. J Dent Oral Hyg. 2010;2(2):19-22.
- 8. Ehrmann E, Messer H, Adams G. The Relationship of Intracanal Medicaments to Postoperative Pain in Endodontics. Int Endod J. 2003;36:868-75.
- 9. Alves Vde O. Endodontic flare-ups: a prospective study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010;110(5):e68-72.
- 10. Tsesis I, Faivishevsky V, Fuss Z, Zukerman O. Flare-ups after endodontic treatment: a metaanalysis of literature. J Endod. 2008;34(10):1177-81.
- 11. Jayakodi H, Kailasam S, Kumaravadivel K, Thangavelu B, Mathew S. Clinical and pharmacological management of endodontic flare-up. J Pharm Bioallied Sci. 2012;4(Suppl 2):S294-8.
- 12. McGurkin-Smith R, Trope M, Caplan D, Sigurdsson A. Reduction of intracanal bacteria using GT rotary instrumentation, 5.25% NaOCl, EDTA, and Ca(OH)2. J Endod. 2005;31(5):359-63.
- 13. Siqueira JF, Jr., Rocas IN, Paiva SS, Guimaraes-Pinto T, Magalhaes KM, Lima KC. Bacteriologic investigation of the effects of sodium hypochlorite and chlorhexidine during the endodontic treatment of teeth with apical periodontitis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007;104(1):122-30.
- 14. Sjogren U, Figdor D, Spangberg L, Sundqvist G. The antimicrobial effect of calcium hydroxide as a short-term intracanal dressing. Int Endod J. 1991;24(3):119-25.
- 15. Siqueira JF, Jr., Magalhaes KM, Rocas IN. Bacterial reduction in infected root canals treated with 2.5% NaOCl as an irrigant and calcium hydroxide/camphorated paramonochlorophenol paste as an intracanal dressing. J Endod. 2007;33(6):667-72.
- 16. Walton RE. Intracanal medicaments. Dent Clin North Am. 1984;28(4):783-96.
- 17. Kim D, Kim E. Antimicrobial effect of calcium hydroxide as an intracanal medicament in root canal treatment: a literature review Part II. in vivo studies. Restor Dent Endod. 2015;40(2):97-103.
- 18. Sundqvist G, Figdor D, Persson S, Sjogren U. Microbiologic analysis of teeth with failed endodontic treatment and the outcome of conservative re-treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998;85(1):86-93.
- 19. Chen BK, George R, Walsh LJ. Discoloration of roots caused by residual endodontic intracanal medicaments. ScientificWorldJournal. 2014;2014:404676.
- 20. Ramos IF, Biz MT, Paulino N, Scremin A, Della Bona A, Barletta FB, et al. Histopathological analysis of corticosteroid-antibiotic preparation and propolis paste formulation as intracanal medication after pulpectomy: an in vivo study. J Appl Oral Sci. 2012;20(1):50-6.
- 21. Jain P, Ranjan M. Role of Herbs in Intracanal Medicaments. Int J Pharm Bio Sci. 2014;5 (3):126-31.

- 22. Yaduka P, Sharma S. Novel Intracanal Medicaments and its Future Scope. Int J Pharm Bio Sci. 2014;4(3):65-9.
- 23. S VK. Propolis in dentistry and oral cancer management. N Am J Med Sci. 2014;6(6):250-9.
- 24. Saha S, Nair R, Asrani H. Comparative Evaluation of Propolis, Metronidazole with Chlorhexidine, Calcium Hydroxide and Curcuma Longa Extract as Intracanal Medicament Against E.faecalis- An Invitro Study. J Clin Diagn Res. 2015;9(11):Zc19-21.
- 25. Shrivastava R, Rai VK, Kumar A, Sinha S, Tripathi P, Gupta K, et al. An in vitro Comparison of Endodontic Medicaments Propolis and Calcium Hydroxide alone and in Combination with Ciprofloxacin and Moxifloxacin against Enterococcus Faecalis. J Contemp Dent Pract. 2015;16(5):394-

9.

- 26. Ferreira FB, Torres SA, Rosa OP, Ferreira CM, Garcia RB, Marcucci MC, et al. Antimicrobial effect of propolis and other substances against selected endodontic pathogens. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007;104(5):709-16.
- 27. Mirzoeva O, Grishanin R, Calder P. Antimicrobial action of propolis and some of its components: the effects on growth, membrane potential and motility of bacteria. Microbiolo Research. 1997;152(3):239-46.
- 28. Neiva K, Catalfamo D, Holliday S, Wallet S, Pileggi R. Propolis decreases lipopolysaccharideinduced inflammatory mediators in pulp cells and osteoclasts. Dent Traumatol. 2014;30:362-7.
- 29. Silvani S, Spettoli E, Stacul F, Tosti A. Contact dermatitis in psoriasis due to propolis. Contact Dermatitis. 1997;37(1):48-9.
- 30. Budimir V, Brailo V, Alajbeg I, Vucicevic Boras V, Budimir J. Allergic contact cheilitis and perioral dermatitis caused by propolis: case report. Acta Dermatovenerol Croat. 2012;20(3):187-90.
- 31. Cho E, Lee JD, Cho SH. Systemic contact dermatitis from propolis ingestion. Ann Dermatol. 2011;23(1):85-8.
- 32. Abbott PV, Hume WR, Heithersay GS. Effects of combining Ledermix and calcium hydroxide pastes on the diffusion of corticosteroid and tetracycline through human tooth roots in vitro. Endod Dent Traumatol. 1989;5(4):188-92.
- 33. Robert GH, Liewehr FR, Buxton TB, McPherson JC, 3rd. Apical diffusion of calcium hydroxide in an in vitro model. J Endod. 2005;31(1):57-60.
- 34. Rehman K, Saunders WP, Foye RH, Sharkey SW. Calcium ion diffusion from calcium hydroxide-containing materials in endodontically-treated teeth: an in vitro study. Int Endod J. 1996;29(4):271-9.
- 35. Montero JC, Mori GG. Assessment of ion diffusion from a calcium hydroxide-propolis paste through dentin. Braz Oral Res. 2012;26(4):318-22.
- 36. Raheja J, Tewari S, Tewari S, Duhan J. Evaluation of efficacy of chlorhexidine intracanal medicament on the periodontal healing of concomitant endodontic-periodontal lesions without communication: an interventional study. J Periodontol. 2014;85(8):1019-26.
- 37. Silva AR, Santos EB, Pinto SC, Gomes JC, Vaz IP, Carvalho MF. Antimicrobial effect and transdentinal diffusion of new intracanal formulations containing nitrofurantoin or doxycycline. Braz Dent J. 2014;25(5):425-9.
- 38. Attia DA, Farag AM, Afifi IK, Darrag AM. Antimicrobial effect of different intracanal medications on various microorganisms. Tanta Dent J. 2015;12(1):41-7.
- 39. Huang S, Zhang C-P, Wang K, Li GQ, Hu F-L. Recent advances in the chemical composition of propolis. Molecules. 2014;19(12):19610-32.
- 40. Tang G, Samaranayake L, Yip HK. Molecular evaluation of residual endodontic microorganisms after instrumentation, irrigation and medication with either calcium hydroxide or Septomixine. Oral Dis. 2004;10(6):389-97.

- 41. Athanassiadis B, Abbott P, Walsh LJ. The use of calcium hydroxide, antibiotics and biocides as antimicrobial medicaments in endodontics. Aust Dent J. 2007;52(s1):S64-S82.
- 42. Gomes B, Souza S, Ferraz C, Teixeira F, Zaia A, Valdrighi L, et al. Effectiveness of 2% chlorhexidine gel and calcium hydroxide against Enterococcus faecalis in bovine root dentine in vitro. Int Endod J. 2003;36(4):267-75.
- 43. Chong B, Ford TP. The role of intracanal medication in root canal treatment. Int Endod J. 1992;25(2):97-106.
- 44. Kikuchi I, Wadachi R, Yoshioka T, Okiji T, Kobayashi C, Suda H. An experimental study on the vasoconstriction effect of calcium hydroxide using rat mesentery. Aust Endod J. 2003;29(3):116-9.
- 45. Grossman LLI, Oliet S, Del Río CE. Endodontic practice. 11th ed. Philadelphia: Lea & Febiger; 1988. 228-33 p.
- 46. Abbott PV. Medicaments: aids to success in endodontics. Part 1. A review of the literature. Aust Dent J. 1990;35(5):438-48.
- 47. Walton RE, Holton IF, Michelich R. Calcium hydroxide as an intracanal medication: effect on posttreatment pain. J Endod. 2003;29(10):627-9.
- 48. Anjaneyulu K, Nivedhitha MS. Influence of calcium hydroxide on the post-treatment pain in Endodontics: A systematic review. J Conserv Dent. 2014;17(3):200.
- 49. Singh RD, Khatter R, Bal RK, Bal C. Intracanal medications versus placebo in reducing postoperative endodontic pain—a double—blind randomized clinical trial. Braz Dent J. 2013;24(1):25-

9.

- 50. QUADIR F, AMIN F, SHAHBAZ U. COMPARISON OF INTRACANAL MEDICATIONS FOR THE ASSESSMENT OF PAIN AFTER ROOT CANAL TREATMENT. Pakistan Oral & Dental Journal. 2015;35(2).
- 51. Mello BC, Hubinger MD. Antioxidant activity and polyphenol contents in Brazilian green propolis extracts prepared with the use of ethanol and water as solvents in different pH values. Int J Food Sci Tech. 2012;47(12):2510-8.
- 52. Li Y, Chen M, Xuan H, Hu F. Effects of encapsulated propolis on blood glycemic control, lipid metabolism, and insulin resistance in type 2 diabetes mellitus rats. Evid Based Complement Alternat Med. 2011;2012.
- 53. Zhu W, Chen M, Shou Q, Li Y, Hu F. Biological activities of Chinese propolis and Brazilian propolis on streptozotocin-induced type 1 diabetes mellitus in rats. Evid Based Complement Alternat Med. 2011;2011.
- 54. Zhu W, Li Y-H, Chen M-L, Hu F-L. Protective effects of Chinese and Brazilian propolis treatment against hepatorenal lesion in diabetic rats. Hum Exp Toxicol. 2011;30(9):1246-55.
- 55. Hu F, Hepburn H, Li Y, Chen M, Radloff S, Daya S. Effects of ethanol and water extracts of propolis (bee glue) on acute inflammatory animal models. J Ethnopharmacol. 2005;100(3):276-83. 56. de Castro Ishida VF, Negri G, Salatino A, Bandeira MFC. A new type of Brazilian propolis: Prenylated benzophenones in propolis from Amazon and effects against cariogenic bacteria. Food Chem. 2011;125(3):966-72.
- 57. Ikeno K, Ikeno T, Miyazawa C. Effects of propolis on dental caries in rats. Caries Res. 1991;25(5):347-51.
- 58. Jafarzadeh Kashi TS, Kermanshahi RK, Erfan M, Vahid Dastjerdi E, Rezaei Y, Tabatabaei FS. Evaluating the in-vitro antibacterial effect of Iranian propolis on oral microorganisms. Iran J Pharm Res. 2011:363-8.
- 59. Jeon J-G, Rosalen P, Falsetta M, Koo H. Natural products in caries research: current (limited) knowledge, challenges and future perspective. Caries Res. 2011;45(3):243-63.

- 60. Momen-Beitollahi J, Mansorian A, Esmaili M, Amanlou M, Mohamadnia A, Bahrami N. Antimicrobial effects of propolis extract on the most prevalent oral pathogens: an in vitro study. Majallah i Dandanpizishki (Journal of Islamic Dental Association of Iran). 2009;21(1):Pe33-Pe9, En8.
- 61. Wang K, Ping S, Huang S, Hu L, Xuan H, Zhang C, et al. Molecular mechanisms underlying the in vitro anti-inflammatory effects of a flavonoid-rich ethanol extract from Chinese propolis (poplar type). Evid Based Complement Alternat Med. 2013;2013.
- 62. Xuan H, Zhao J, Miao J, Li Y, Chu Y, Hu F. Effect of Brazilian propolis on human umbilical vein endothelial cell apoptosis. Food Chem Toxicol. 2011;49(1):78-85.
- 63. Xuan H, Zhu R, Li Y, Hu F. Inhibitory effect of chinese propolis on phosphatidylcholinespecific phospholipase C activity in vascular endothelial cells. Evid Based Complement Alternat Med. 2010;2011.
- 64. Bankova V, De Castro S, Marcucci M. Propolis: recent advances in chemistry and plant origin. Apidologie. 2000;31(1):3-15.
- 65. Ito J, Chang F-R, Wang H-K, Park YK, Ikegaki M, Kilgore N, et al. Anti-AIDS agents. 48. 1 Anti-HIV activity of moronic acid derivatives and the new melliferone-related triterpenoid isolated from Brazilian propolis. J Nat Prod. 2001;64(10):1278-81.
- 66. Koo H, Gomes B, Rosalen P, Ambrosano G, Park Y, Cury J. In vitro antimicrobial activity of propolis and Arnica montana against oral pathogens. Arch Oral Biol. 2000;45(2):141-8.
- 67. Feres M, Figueiredo L, Barreto I, Coelho M, Araujo M, Cortelli S. In vitro antimicrobial activity of plant extracts and propolis in saliva samples of healthy and periodontally-involved subjects. J Int Acad Periodontol. 2005;7(3):90-6.
- 68. Tanasiewicz M, Skucha-Nowak M, Dawiec M, Król W, Skaba D, Twardawa H. Influence of hygienic preparations with a 3% content of ethanol extract of brazilian propolis on the state of the oral cavity. Adv Clin Exp Med. 2012;21(1):81-92.
- 69. Pereira EMR, da Silva JLDC, Silva FF, De Luca MP, Lorentz TCM, Santos VR. Clinical evidence of the efficacy of a mouthwash containing propolis for the control of plaque and gingivitis: a phase II study. Evid Based Complement Alternat Med. 2011;2011.
- 70. Schnitzler P, Neuner A, Nolkemper S, Zundel C, Nowack H, Sensch KH, et al. Antiviral activity and mode of action of propolis extracts and selected compounds. Phytother Res. 2010;24(S1):S20S8.
- 71. Özan F, Polat ZA, Er K, Özan Ü, Değer O. Effect of propolis on survival of periodontal ligament cells: new storage media for avulsed teeth. J Endod. 2007;33(5):570-3.
- 72. Gulinelli JL, Panzarini SR, Fattah CMRdS, Poi WR, Sonoda CK, Negri MR, et al. Effect of root surface treatment with propolis and fluoride in delayed tooth replantation in rats. Dent Traumatol. 2008;24(6):651-7.
- 73. Gopikrishna V, Baweja PS, Venkateshbabu N, Thomas T, Kandaswamy D. RETRACTED: Comparison of Coconut Water, Propolis, HBSS, and Milk on PDL Cell Survival. J Endod. 2008;34(5):587-9.
- 74. Magro-Filho O, Carvalho ACPd. Topical effect of propolis in the repair of sulcoplasties by the modified Kazanjian technique. Cytological and clinical evaluation. J Nihon Univ Sch Dent. 1994;36(2):102-11.
- 75. Lopes Rocha R, Miranda Jd, Lima NL, Ferreira FO, Marinho SA, Verli FD. Effect of topical propolis and dexamethasone on the healing of oral surgical wounds. Wound Healing Southern Africa. 2012;5(1):25-30.
- 76. Altan BA, Kara IM, Nalcaci R, Ozan F, Erdogan SM, Ozkut MM, et al. Systemic propolis stimulates new bone formation at the expanded suture: a histomorphometric study. Angle Orthod. 2012;83(2):286-91.
- 77. Sales-Peres SHdC, Carvalho FNd, Marsicano JA, Mattos MC, Pereira JC, Forim MR, et al. Effect of propolis gel on the in vitro reduction of dentin permeability. J Appl Oral Sci. 2011;19(4):31823.

- 78. Ahangari Z, Naseri M, Jalili M, Mansouri Y, Mashhadiabbas F. Torkaman Pharm A. Effect of propolis on dentin regeneration and the potential role of dental pulp stem cell in Guinea Pigs. Cell J. 2012; 13 (4): 2230228. Cell J. 2012;13(4):223.
- 79. Ozório JEV, de Oliveira DA, de Sousa-Neto MD, Perez DEdC. Standardized propolis extract and calcium hydroxide as pulpotomy agents in primary pig teeth. J Dent Child (Chic). 2012;79(2):53-8.
- 80. Parolia A, Kundabala M, Rao N, Acharya S, Agrawal P, Mohan M, et al. A comparative histological analysis of human pulp following direct pulp capping with Propolis, mineral trioxide aggregate and Dycal. Aust Dent J. 2010;55(1):59-64.
- 81. Valera MC, da Rosa JA, Maekawa LE, de Oliveira LD, Carvalho CA, Koga-Ito CY, et al. Action of propolis and medications against Escherichia coli and endotoxin in root canals. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010;110(4):e70-4.
- 82. Mattigatti S, Ratnakar P, Moturi S, Varma S, Rairam S. Antimicrobial effect of conventional root canal medicaments vs propolis against Enterococcus faecalis, Staphylococcus aureus and Candida albicans. J Contemp Dent Pract. 2012;13(3):305-9.
- 83. Kayaoglu G, Omurlu H, Akca G, Gurel M, Gencay O, Sorkun K, et al. Antibacterial activity of Propolis versus conventional endodontic disinfectants against Enterococcus faecalis in infected dentinal tubules. J Endod. 2011;37(3):376-81.
- 84. Awawdeh L, Al-Beitawi M, Hammad M. Effectiveness of propolis and calcium hydroxide as a short-term intracanal medicament against Enterococcus faecalis: a laboratory study. Aust Endod J. 2009;35(2):52-8.
- 85. Madhubala MM, Srinivasan N, Ahamed S. Comparative evaluation of propolis and triantibiotic mixture as an intracanal medicament against Enterococcus faecalis. J Endod. 2011;37(9):1287-9.
- 86. Carbajal Mejía JB. Antimicrobial effects of calcium hydroxide, chlorhexidine, and propolis on Enterococcus faecalis and Candida albicans. J Investig Clin Dent. 2014;5(3):194-200.
- 87. Chua EG, Parolia A, Ahlawat P, Pau A, Amalraj FD. Antifungal effectiveness of various intracanal medicaments against Candida albicans: an ex-vivo study. BMC oral health. 2014;14(1):1.
- 88. Jahromi MZ, Ranjbarian P, Shiravi S. Cytotoxicity evaluation of Iranian propolis and calcium hydroxide on dental pulp fibroblasts. J Dent Res Dent Clin Dent Prospects. 2014;8(3):130.
- 89. Ali AH, Najeh S. In vitro toxicity of propolis in comparison with other primary teeth pulpotomy agents on human fibroblasts. J Investig Clin Dent. 2015.
- 90. Ramos IFdAS, Biz MT, Paulino N, Scremin A, Della Bona Á, Barletta FB, et al. Histopathological analysis of corticosteroid-antibiotic preparation and propolis paste formulation as intracanal medication after pulpectomy: an in vivo study. J Appl Oral Sci. 2012;20(1):50-6.
- 91. Silva FBd, Almeida JMd, Sousa SMGd. Natural medicaments in endodontics: a comparative study of the anti-inflammatory action. Braz Oral Res. 2004;18(2):174-9.
- 92. Neiva KG, Catalfamo DL, Holliday S, Wallet SM, Pileggi R. Propolis decreases lipopolysaccharide-induced inflammatory mediators in pulp cells and osteoclasts. Dent Traumatol. 2014;30(5):362-7.
- 93. Ørstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Dent Traumatol. 1986;2(1):20-34.
- 94. Ehrmann EH, Messer HH, Clark RM. Flare-ups in endodontics and their relationship to various medicaments. Aust Endod J. 2007;33(3):119-30.
- 95. Population explosion: Put an embargo on industrialisation in Karachi. <a href="http://tribunecompk">http://tribunecompk</a>. 6 october 2013.
- 96. Shah SA, Maxood A, Shah SI. Incidence of Endodontic Flare–UPS using either calcium hydroxide or Creosote as intracanal Medicament in Symptomatic teeth. Journal of Khyber College of Dentistry. 2010;1:1.

- 97. Xavier ACC, Martinho FC, Chung A, Oliveira LD, Jorge AO, Valera MC, et al. One-visit versus two-visit root canal treatment: effectiveness in the removal of endotoxins and cultivable bacteria. J Endod. 2013;39(8):959-64.
- 98. Martinho FC, Nascimento GG, Leite FR, Gomes AP, Freitas LF, Camoes IC. Clinical influence of different intracanal medications on Th1-type and Th2-type cytokine responses in apical periodontitis. J Endod. 2015;41(2):169-75.

#### 3.2 – Appendices:

## **VISUAL(PAIN) ANALOGUE SCALE**



On a scale from 0-100(given above), please mark the intensity of pain at different times using the criteria(chart) given on the right side:

- 1) Before start of treatment =
- 2) 04 hours =
- *3) -* 12 hours =
- 4) Day 2 =
- *5)* Day 3 =
- 6) Day 4 =

Patient Serial No. =

- **0-24**=> No pain to mild pain, requires no pain killer.
  - <u>25-49</u>=> Moderate pain requires Ibuprofen, or similar medication for relief.
  - **50-74**=> Severe pain not relieved by above medication necessitating use of narcotic analgesics such as Codeincontaining preparations.

**75-100**=> Extreme pain not relieved by any measures taken.

Chart: criteria for assessing the pain severity

#### **Informed Consent Form**



# EFFECT OF PROPOLIS PASTE AS INTRACANAL MEDICAMENT ON POST-ENDODONTIC PAIN: A DOUBLE BLIND RANDOMIZED CLINICAL TRIAL

| PRINCIPAL RESEARCHER | WITNESS | CSS CONTACT DETAILS |
|----------------------|----------------------------|---------------------|
| DR. JUZER SHABBIR | Dr.juzer.shabbir@gmail.com | |

- I consent to participate in the project named above which is taking place in Doctor Ishrat-ul-ibad khan Institute of Oral Health Sciences. The particulars of participation have been explained to me.
- I acknowledge that:
  - (a) The possible effects of the use of these data have been explained to me to my satisfaction
  - (b) The project is for the purpose of research for assessment in higher education.
- I understand that:
  - (a) My identity will not be revealed in any report based on this project. (b) This consent form and data I supply will be kept in confidence by the researchers.

#### Information consent (choose one): YES NO

- I authorize the researchers to record and analyze data for the stated purposes of the project.
- I have been informed that the confidentiality of the information I provide will be safeguarded subject to any legal requirements.

| | | T |
|------|-----|-----|
| Name | Age | Sex |

Thank you.